CLINICAL TRIAL: NCT00016497
Title: Adenoidectomy for Otitis Media in 2-3 Year Old Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: NIDCD1RO1DC035-04
Record Dates: First submitted 2001-05-10; First posted 2001-05-14 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Otitis Media With Effusion
Keywords: otitis media with effusion; children; tympanostomy tubes; adenoidectomy
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Adenoidectomy

INTERVENTIONS:
Procedure: bilateral myringotomy
Procedure: bilateral myringotomy and tubes
Procedure: adenoidectomy

SUMMARY:
The purpose of this study is to evaluate the efficacy of three different surgical treatments (1. Bilateral myringotomy and tube insertion (M&T); 2. Adenoidectomy and bilateral myringotomy (A&T); 3. Adenoidectomy with myringotomy and tympanostomy tube insertion (A-M&T)) in reducing subsequent episodes of middle ear disease and hearing loss caused by the fluid in the middle ear in children aged 24-47 months. The fluid in the middle ear is of at least three months' duration and unresponsive to standardized, recent antimicrobial treatment. The children are assigned to one of the three surgical treatments. After surgery, they are followed with examinations monthly and at the time of intercurrent infections for three years.

DETAILED DESCRIPTION:
The specific aim of this study is to compare, by means of a randomized clinical trial, the efficacy of three surgical treatment combinations: adenoidectomy with myringotomy (A-M), adenoidectomy with myringotomy and tympanostomy tube insertion (A-M&T), and M&T alone, in reducing subsequent middle ear disease in children aged 24-47 months with otitis media with effusion (OME) of at least 3 months' duration unresponsive to standardized, recent antimicrobial treatment. The children are randomly assigned to one of three treatment arms: 1. M&T; 2. A-M; and 3. A-M&T. Subjects are be stratified according to: 1. age; 2. nasal obstruction; and 3. previous tubes. All subjects are scheduled for surgery according to assignment within 4 weeks after entry. The first post-operative visit takes place 2 weeks after surgery, and a complete examination of the ears, nose, and throat (ENT exam) including pneumatic otoscopy, tympanometry and audiometry is performed. Subjects are followed with monthly evaluations (ENT-exam, pneumatic otoscopy, tympanometry) for three years. Audiometry is performed every 6 months. All subjects are evaluated at any time while still enrolled in the study if signs and symptoms of URI, acute otitis media (AOM, including otorrhea), or OME occur and are treated appropriately. Subjects who develop OME for 4 months bilaterally or 6 months unilaterally have M&T and continue to be followed in the study. The primary outcome measure will be percentage of time with middle ear effusion (MEE). Episodes of AOM, otorrhea, and OME, time to first recurrence, and number of surgical procedures will be compared between the three treatment groups. Treatment failures, complications and sequelae of treatments will also be recorded and compared among the three treatment groups.

ELIGIBILITY:
* Males and females between 24 and 47 months of age, in good general health.
* Asymptomatic otitis media with effusion bilaterally for a minimum of 3 consecutive months.
* At least one 10-day course of a broad-spectrum antimicrobial agent in the last month.

Ages: 24 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1997-02; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Margaretha L Casselbrant, Principal Investigator — University of Pittsburgh
Locations (1):
- Ear, Nose, and Throat Research Center, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States